CLINICAL TRIAL: NCT05544656
Title: The Prognostic Value of Biomarkers and the Effect of Tolperisone in Acute Low Back Pain -BETA. A Phase 3 Investigator Initiated Study
Brief Title: The Prognostic Value of Biomarkers and the Effect of Tolperisone in Acute Low Back Pain and Sciatic Pain "BETA"
Acronym: BETA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: National Research Develpment and Innovation Fund, Hungary (Unknown); MEDITOP Pharmaceutical LTD, Hungary (Unknown)
Responsible Party: Principal Investigator, Daniel Bereczki, Professor of neurology, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOWBACK-SE-01
Record Dates: First submitted 2022-08-08; First posted 2022-09-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
Keywords: back pain; sciatic pain; biomarkers
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Tolperisone

STUDY DESIGN:
Intervention Model Description: Single center, randomized double blind study. Randomization is done separately for those with and those without radicular signs.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization is done by non-transparent (opaque) sequentially numbered envelopes, prepared independently from the trial site. The number on the envelope corresponds to the number on the boxes of the trial medication (tolperisone or matching placebo). The envelopes can be opened only at the end of the trial, or in case of emergency. No interim analysis is planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tolperisone (Experimental): Tolperisone 3 times 150 mg daily, i.e. a daily dose of 450 mg. Treatment lasts for 14 days
  Interventions: Drug: Tolperisone Hydrochloride
- Placebo (Placebo Comparator): Matching placebo 3 times daily. Treatment lasts for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolperisone Hydrochloride — Tolperisone Hydrochloride tablets of 150 mg, administered three times a day
  Other Names: EV product code: PRD4558977, miderizone tablet, ATC:M03BX04
  Arms: Tolperisone
Drug: Placebo — matching placebo administered three times a day
  Arms: Placebo

SUMMARY:
The main purpose of the trial is to identify biomarkers from the blood as well as electrophysiologic and morphometric features (chemical, electrophysiologic and ultrasound biomarkers) that reflect the intensity of pain and/or foretell the efficacy of pharmacological (non-surgical) treatment in patients with acute low back pain.

DETAILED DESCRIPTION:
The investigators include patients aged 18-80 years with acute (less than 1-month) low back pain with or without radicular signs, who do not have severe diseases (abscess, tumor, etc) in the background, already had CT or MRI scan during routine workup, and who have given written consent to participate in the study. Exclusion criteria are pregnancy, hypersensitivity to tolperisone in the history, severe liver or kidney disease, other severe diseases (abscess, tumor, etc) in the background of pain. The patients will be given 3 times daily 150 mg tolperisone or placebo in addition to standard therapy in a randomized double-blind design. Treatment will last for 14 days and a final follow-up is performed at 21 days. Clinical condition and biomarkers will be tested before treatment and at 14 days. Patients fill in a diary on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pain-free volunteers (n=30) outside of the randomized study, will participate to establish normal values of blood biomarkers.

Exclusion Criteria:

* pain, inflammation,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the level of biomarkers by the end of the treatment period compared to the pretreatment values. | 14 days
  Changes in the values of blood biomarkers (nociceptin/orphanin FQ, Met-Enkephalin-Arg6-Phe7 (MEAP), pro-inflammatory cytokines (IL-1β, IL-6, IL-2, IL-8, IL-12, IL-33, CCL3, CXCL1, CCR5, és TNF-α), anti-inflammatory cytokines (IL-10 and IL-4), monocyte chemoattractant protein-1 (MCP-1), macrophage inflammatory proteins-1b (MIP-1b), platelet-derived growth factor (PDGF AA), vascular endothelial growth factor (VEGF), GM-CSF=granulocyte-macrophage colony-stimulating factor, CGRP (calcitonin gene related peptide), substance P, noradrenalin (norepinephrine), in electrophysiologic markers (quantitative electromyography with surface electrodes in the paravertebral muscles in prone and standing position) and ultrasound markers (bilateral measurements of cross sectional area and antero-posterior diameter of paravertebral muscles in prone and standing position)
Patient reported change in pain features | daily for 14 days
  Self evaluation of pain by the patient on a visual scale from zero (no pain at all) to 10 (the most severe pain the patient can imagine)

SECONDARY OUTCOMES:
Change in the level of biomarkers enlisted in Primary Outcome 1 in the subgroup of those with ceased or greatly reduced pain | 14 days
  Subgroup analysis of the change in biomarkers restricted to those with ceased or greatly reduced pain
Change in the intensity of pain by the end of the treatment period | 14 days
  Self evaluation of pain by the patient on a visual scale from zero (no pain at all) to 10 (the most severe pain the patient can imagine)
Change in the level of biomarkers enlisted in Primary Outcome 1 by the end of the treatment period in the tolperisone group | 14 days
  Subgroup analysis of changes in blood, electrophysiological and ultrasound biomarkers by 14 days in the tolperisone group
Change in the level of paravertebral muscle contraction by the end of the treatment period | 14 days
  Analysis restricted to the electrophysiological and ultrasound biomarkers enlisted in Primary Outcome 1
Predictive value of the initial levels of biomarkers enlisted in Primary Outcome 1 | 14 days
  Evaluation of the association of the initial biomarker values enlisted in Primary Outcome 1 with the 14-day pain features
Global impression of change by the patient | 14 days
  Patient self evaluation of changes by the end of treatment on a 6-grade scale (has become symptom-free; major improvement; minor improvement; no change; minor worsening; major worsening)
Global clinical impression of change (GCI) by the investigator | 14 days
  Subjective evaluation of changes by the end of treatment on a 6-grade scale by the investigator (has become symptom-free; major improvement; minor improvement; no change; minor worsening; major worsening)
Number of participants with treatment-related adverse events | 21 days (14 days treatment plus 7 days post-treatment)
  Any adverse events reported during the 14 days of treatment and the 7-day post-treatment period

OTHER OUTCOMES:
Patient reported sleep quality | Daily from 1-14 days
  Changes in sleep quality reported in patient diary on a 4-grade scale (1: undisturbed sleep; 2: woke up once due to pain; 3: woke up more than once due to pain; 4: could not sleep at all due to pain).
Fingertip-to-floor distance | 14 days
  The patient is asked to bend forward and attempt to reach for the floor with their fingertips. The distance between the patient's right long finger and the floor is measured using a standard measuring tape in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bereczki, MD, POhD,DSc, Principal Investigator — Semmelweis University
Locations (1):
- Department of Neurology, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
After trial completion the investigators will be ready to share data with other researchers based on reasonable request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Infinite afer trial completion
Access Criteria: request should be discussed by email of the principal investigator